CLINICAL TRIAL: NCT04313504
Title: An Open-label, Phase II Study Evaluating the Efficacy of Niraparib and Dostarlimab (TSR-042) in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Study Evaluating the Efficacy of Niraparib and Dostarlimab (TSR-042) in Recurrent/Metastatic HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trisha Wise-Draper (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-19-03
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib & Dostarlimab (Experimental): Niraparib starting on Day 0. Niraparib will be administered as continuous daily dose, orally 200 or 300 mg.
  Dostarlimab IV administered via a 30-minute infusion on Day 1 of every 21 day cycle. 500mg for first 4 doses followed by 1000 mg every 6 weeks.
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — Niraparib & Dostarlimab combination
  Other Names: ZEJULA
Drug: Dostarlimab — Niraparib & Dostarlimab combination
  Other Names: TSR-042

SUMMARY:
The purpose of this study is to determine the best overall response of the combination of dostarlimab and niraparib in patients with recurrent and/or metastatic HNSCC patients.

DETAILED DESCRIPTION:
Recurrent and/or metastatic HNSCC patients will be treated with combination of the PD-1 inhibitor (dostarlimab) and PARPi (niraparib) concurrently and ORR, PFS and OS will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically, cytologically, or radiographically confirmed recurrent or metastatic non cutaneous HNSCC for which there are no surgical or radiation curative options.
* ECOG performance status ≤2
* Patients must be able to swallow pills

Exclusion Criteria:

* Nasopharyngeal and salivary gland tumors
* Patients who have not recovered from adverse events due to prior anti-cancer therapy with the exception of alopecia
* Prior exposure to both immunotherapy drugs (PD-1, PDL-1, CTLA-4 inhibitors) and PARP inhibitors. Single exposure to either immunotherapy or PARP inhibitors is allowable.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to niraparib or dostarlimab.
* Patients with uncontrolled intercurrent illness.
* Requirement of any use of steroids greater than the equivalent of 10mg prednisone daily is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 8 weeks
  Measured by assessing best overall response using RECIST 1.1 in subjects in recurrent and/or metastatic HNSCC patients receiving combination of niraparib and dostarlimab.

SECONDARY OUTCOMES:
Rate of all Adverse Events | 30 days after completion of treatment
  As determined by CTCAE v5.0 in subjects with recurrent and/or metastatic HNSCC receiving combination of niraparib and dostarlimab.
Progression Free Survival | 1 and 3 years
  Measured using Kaplan Meier Curves from time of treatment start until time of progression
Overall Survival | 5 years
  Measured using Kaplan Meier Curves from diagnosis until time of death

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No